CLINICAL TRIAL: NCT01723124
Title: Comparison of Breast Cancer Detection Rate for Prevalent Screen Low-dose Molecular Breast Imaging and Incident Biennial Screen Low-dose Molecular Breast Imaging in Women With Mammographically Dense Breasts
Brief Title: Low-dose Molecular Breast Imaging: Comparison of Breast Cancer Detection Rate at Initial Screening and Two-year Follow-up
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dose specified in protocol was not adequate to achieve optimal resolution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Rhodes, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-004322
Record Dates: First submitted 2012-07-24; First posted 2012-11-07 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Dense breast tissue; breast cancer screening; molecular breast imaging; breast cancer; breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Molecular Breast Imaging (Experimental): Molecular Breast Imaging (MBI) utilizes small high resolution gamma camera detectors in a dual-detector configuration to image the breast following the administration of a radiopharmaceutical that accumulates preferentially in breast tumors.
  Interventions: Procedure: Molecular Breast Imaging

INTERVENTIONS:
Procedure: Molecular Breast Imaging — Molecular Breast Imaging (MBI) utilizes small high resolution gamma camera detectors in a dual-detector configuration to image the breast following the administration of a radiopharmaceutical that accumulates preferentially in breast tumors.

SUMMARY:
The purpose of this research is to evaluate whether repeating a screening Molecular Breast Imaging (MBI) study two years after an initial screening MBI study further improves breast cancer detection in women with dense breast tissue.

ELIGIBILITY:
Inclusion Criteria:

- Past prior screening mammogram within the previous 11-24 months interpreted as heterogeneously dense or extremely dense and negative or benign [Breast Imaging Reporting and Data System (BI-RADS) Category 1 or 2]

Exclusion Criteria:

Subjects will be excluded if they:

* Are unable to understand and sign the consent form
* Are pregnant or lactating
* Are physically unable to sit upright and still for 40 minutes
* Have self-reported signs or symptoms that may suggest breast cancer (palpable mass, bloody nipple discharge, axillary mass, etc.)
* Have had needle biopsy within 3 months, or breast surgery or radiation within 1 year prior to the study
* Are currently receiving chemotherapy or tamoxifen, raloxifene, or an aromatase inhibitor for adjuvant therapy or chemoprevention
* Have undergone bilateral mastectomy
* Have had a prior MBI within 20 months of scheduled study MBI.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Molecular Breast Imaging (MBI) scan | Performed at Year 0 of study
  The Year 0 MBI will be interpreted in isolation, with the radiologist blinded to Year 0 mammogram results and all relevant clinical information.

SECONDARY OUTCOMES:
Molecular Breast Imaging (MBI) scan | Performed at Year 2 of study
  The Year 2 MBI will be interpreted in comparison with the Year 0 MBI but in isolation from the Year 2 mammogram.

OTHER OUTCOMES:
Comparison of breast cancer detection rate for Year 0 and Year 2. | Year 2 of study
  The breast cancer detection rate for Year 0 and Year 2 MBI will be compared to each other and to the breast cancer detection rates for the screening mammograms performed in Year 0 and Year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rhodes, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes DJ, Hruska CB, Phillips SW, Whaley DH, O'Connor MK. Dedicated dual-head gamma imaging for breast cancer screening in women with mammographically dense breasts. Radiology. 2011 Jan;258(1):106-18. doi: 10.1148/radiol.10100625. Epub 2010 Nov 2. PMID 21045179
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0